CLINICAL TRIAL: NCT06313684
Title: Comprehensive Hybrid Cardiac Rehabilitation Trial to Assess Impact on Heart Failure Patients
Brief Title: Comprehensive Hybrid Cardiac Rehabilitation Trial on Heart Failure
Acronym: COCREATIONHF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Collaborators: University of Chile (Other)
Responsible Party: Principal Investigator, Pamela Serón, Principal Investigator, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fondecyt 1230787
Record Dates: First submitted 2024-03-04; First posted 2024-03-15 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III
Keywords: cardiac rehabilitation; heart failure; exercise
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Psychiatric Rehabilitation; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comprehensive Hybrid Cardiac Rehabilitation (Experimental): The 24-week Cardiac Rehabilitation intervention will include evaluation, medical and nurse management, aerobic interval training, resistance exercise, psychosocial support, and education. These will initially be delivered in a health center, transitioning to home in 4 stages.
  Interventions: Other: Comprehensive Initial Assessment; Other: Continuous evaluation; Other: Interval Exercise; Behavioral: Psychosocial support; Other: Diet management; Other: Resistance exercise
- Exercise and center-based Cardiac Rehabilitation (Active Comparator): Cardiac rehabilitation with face-to-face continuous aerobic exercise sessions and resistance exercises.
  Interventions: Other: Resistance exercise; Other: Continuous exercise; Other: Initial Assessment

INTERVENTIONS:
Other: Comprehensive Initial Assessment — Initial Assessment includes all those necessary to prescribe exercise training, as well as dietary and adherence promotion interventions.
  * Functional capacity with 6MWT
  * Assessment of skeletal muscle strength, flexibility, and balance.
  * Assessment of function
  * Assessment of dietary habits
  * Assessment of self-efficacy and barriers to CR adherence.
  * Screening for depression.
  Arms: Comprehensive Hybrid Cardiac Rehabilitation
Other: Continuous evaluation — Evaluations during the course of the program will be carried out to inform the progression through the CR stages, the intensity of training and education needs.
  Arms: Comprehensive Hybrid Cardiac Rehabilitation
Other: Interval Exercise — High-intensity interval training prescribed by physical therapist:
  * According to an adapted Wisloff protocol.
  * Borg scale to monitor intensity.
  * Training 3 times per week.
  Arms: Comprehensive Hybrid Cardiac Rehabilitation
Behavioral: Psychosocial support — Based on social-cognitive theory, with self-efficacy as a focus:
  * Face-to-face sessions in the first stage of the program: Education, self-monitoring and motivational interview.
  * Face-to-face session in the second stage of the program: promoting behavior changes by self-control and self-monitoring
  * Regular communication with patients will be supported by the use of mobile devices during the third and fourth stages of program.
  Arms: Comprehensive Hybrid Cardiac Rehabilitation
Other: Diet management — A dietary plan supported by a nutritionist will be made together with the patient.
  Arms: Comprehensive Hybrid Cardiac Rehabilitation
Other: Resistance exercise — Resistance exercises:
  * With TheraBand.
  * Intensity according to the perceived exertion scale
  * Twice a week.
Other: Continuous exercise — Moderate-intensity continuous exercise prescribed by physical therapist :
  * The intensity will be moderate, as tolerated
  * Borg scale to monitor intensity.
  * Frequency of training of 1 to 3 times per week, until completed 20 sessions in 10-12 weeks.
  Arms: Exercise and center-based Cardiac Rehabilitation
Other: Initial Assessment — Includes all those necessary to plan exercise training, as usual:
  * Functional capacity with 6MWT.
  * Assessment of skeletal muscle strength.
  Arms: Exercise and center-based Cardiac Rehabilitation

SUMMARY:
CO-CREATION-HF aims to evaluate the effectiveness of a comprehensive and hybrid cardiac rehabilitation model compared to supervised exercise alone.

DETAILED DESCRIPTION:
Comprehensive, hybrid cardiac rehabilitation (CR) models have been scantly investigated in heart failure (HF) populations, particularly in low-resource settings.

A 2 parallel-arm, multi-center randomized clinical superiority trial will be conducted with blinded outcome assessment. 152 HF patients (NYHA class II or III) will be recruited consecutively, and randomly assigned. The experimental intervention will include evaluation, medical and nurse management, aerobic interval training, resistance exercise, psychosocial support, and education. These will initially be delivered in a center, transitioning to home in 4 stages. Participants in the control arm will receive face-to-face continuous aerobic exercise sessions and resistance exercises. The main outcomes are cardiorespiratory fitness, functional capacity, and quality of life. These will be measured at baseline, end of intervention, and 12-month follow-up.

The pragmatic, comprehensive hybrid CR model could be implemented more broadly if superiority is demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with HF of New York Heart Association functional class II or III.
* Meets HF diagnostic criteria of Guidelines
* On optimal tolerated medical therapy.
* Deemed by the treating physician as stable for at least 1 month.
* Able to attend the health center three times a week for the first month, and twice a week for the 2nd and 3rd months
* Owns a mobile phone
* Patient consents to participate in the study by signing an informed consent form.

Exclusion Criteria:

* Chronic kidney disease with glomerular filtration rate < 20 mL/min.
* Decompensated thyroid disease.
* End-stage liver failure or Child-Pugh C.
* Cardiac device or cardiac surgery in the previous month or planned in the next 3 months.
* Patients with dyspnea predominantly of non-cardiac cause (e.g. COPD).
* Atrial fibrillation with a heart rate greater than 90 beats per minute at rest.
* Active neoplasm with life expectancy <2 years.
* Inclusion in another interventional study.
* Explicit contraindications to performing exercise.
* Comorbidities that preclude the patient from engaging in a CR program.
* Musculoskeletal or neurological disease that precludes the patient from performing exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | Baseline, 6 months and 12 months.
  Will be assessed during a symptom-limited cardiopulmonary exercise test using an individualized gradual incremental ramp test designed to obtain oxygen consumption (VO2max).
Functional capacity | Baseline, 6 months and 12 months.
  Will be assessed by the six-minute walk test (6MWT)
Health Related Quality of Life | Baseline, 6 months and 12 months.
  Will be evaluated with the Minnesota Living with Heart Failure Questionnaire (MLHFQ). This questionnaire has 21 questions, which are answered on a scale of 1 to 5. The score of the questionnaire is obtained by the sum of the answers to the 21 questions, the higher the score, the worse the quality of life.

SECONDARY OUTCOMES:
Program adherence and completion | 6 months
  Program adherence is defined as the percentage of total prescribed sessions completed. For home-based activities, the percentage of activities carried out at home of the prescribed ones will be computed.
Concentration of Pro-B-type Natriuretic Peptide | Baseline, 6 months and 12 months.
  Biomarker with prognostic utility. When it is higher than 1000 pg/mL, there is a higher probability of having events such as hospitalizations.
Functioning | Baseline, 6 months and 12 months.
  Defined as the ability to perform basic, instrumental and advanced activities of daily living. It will be measured with the Activities of Daily Living Questionnaire - Technology (ADLQ-T). This questionnaire evaluates 7 areas: self-care (6 items), home care and management (6 items), work and recreation (4 items), shopping and money (3 items), travel (3), communication (5 items) and technology (5 items). Each item has a score, where 0 is no problem for the activity up to 3 indicating that he/she cannot perform the activity. The functional deficit is calculated for each area and for the overall questionnaire with the sum of all scores, divided by 3 and then multiplied by the total number of items answered. A higher score indicates greater impairment of ADLs.
Mortality and Hospital admission | 12 months
  Will be measured as a composite outcome. It will be measured as a composite outcome. An adjudicating committee will confirm the events that will be expressed as the number of participants hospitalized or dead and their respective causes. All-cause and HF-specific mortality and hospitalization will be differentiated.
Upper-body muscle strength | Baseline, 6 months and 12 months.
  Will be assessed through grip strength performed with a Jamar® Plus+ electronic handheld dynamometer. the result shall be expressed in kilograms.
Lower-body muscle strength | Baseline, 6 months and 12 months.
  Will be assessed through the chair stand test, with the participant in a seated position in a chair. From this position, they will be directed to rise fully and return to the starting position as many times as possible over 30 seconds. The number of repetitions achieved will be recorded
Cost | 6 months
  Will be assessed through micro-costing from the health care system perspective. Also out-of-pocket spending by patients will be costed

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Seron, PhD, Principal Investigator — Universidad de La Frontera
Locations (4):
- Chile (4):
  - Complejo Hospitalario San José, Santiago
  - Hospital Clínico Universidad de Chile, Santiago
  - Hospital San Borja Arriarán, Santiago
  - Universidad de La Frontera, Temuco

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the main results article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 6 months following main results article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee.
  For individual participant data meta-analysis. Proposals should be directed to Principal Investigator. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Seron P, Gomez-Perez D, Opazo-Diaz E, Oliveros MJ, Contreras MF, Salinas A, Andrade-Mayorga O, Marzuca-Nassr GN, Saavedra K, Espejo C, Munoz S, Lanas F, Grace SL. CO-CREATION-HF protocol: clinical trial to evaluate the impact of a comprehensive and hybrid cardiac rehabilitation model on patients with heart failure. Front Cardiovasc Med. 2024 Nov 14;11:1427544. doi: 10.3389/fcvm.2024.1427544. eCollection 2024. PMID 39610971